CLINICAL TRIAL: NCT04481568
Title: Reducing Behavioral and Psychological Symptoms of Dementia (BPSD) for Acutely-Ill Persons With Alzheimers Disease and Related Dementias Via Patient Engagement Specialists
Brief Title: Reducing Behavioral and Psychological Symptoms of Dementia: Family Caregivers (Aim 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 19-0800-FIMR-1; 1R21NR018500-01 (NIH)
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Alzheimer's Disease and Related Dementias
Keywords: Behavioral and Psychological Symptoms of Dementia; Alzheimer's Disease and Related Dementias; Hospitalization
MeSH Terms: conditions — Alzheimer Disease; Behavior

STUDY DESIGN:
Intervention Model Description: Nonrandom preliminary efficacy trial comparing 2 groups, intervention and control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The PES-4-BPSD Model (Experimental): The intervention arm consists of PES and nurse assistants who work on the intervention unit which consists of: I. Cohorting of patients with cognitive impairment AND past or present indication of BPSD, acutely admitted to the medicine or telemetry service, are cohorted on a 10-bed medical unit. II. PES staff: mental health assistants with high school level education, who receive training in de-escalation and crisis prevention techniques and provide direct personal care to psychiatric patients. On the intervention unit, these PES purposefully engage patients with BPSD. III. Staff Support: The PI will hold monthly 20 minute group sessions to reinforce training and discuss challenging patient behaviors; meant to improve the attitude and empathy of HCGs towards patients. IV. Staff Training (please refer to NCT# 04179721 for more details on staff support and training).
  Interventions: Behavioral: PES-4-BPSD Model
- The attention control condition (Active Comparator): The attention control condition will consist of a 40-bed medicine unit, staffed with 39 nurses (1:6 ratio) and 26 nursing assistants (1:8 ratio), that primarily cohorts older patients with geriatric syndromes.
  Interventions: Behavioral: The attention control condition

INTERVENTIONS:
Behavioral: PES-4-BPSD Model — We will conduct a non-randomized preliminary efficacy trial, enrolling N=158 patients (79 control and 79 intervention). The primary outcome will be presence of BPSD as measured by a patient's total score on the Neuropsychiatric Inventory-Questionnaire (NPI-Q) during hospitalization. A multi-modal approach (including chart review and HCG questionnaires) will be used to determine the presence and severity of BPSD.
  Arms: The PES-4-BPSD Model
Behavioral: The attention control condition — On this unit, the management of patients who display BPSD is performed by nurse assistants, rather than PES. Therefore, in order to test the added layer of PES staff, the nurse assistants on the control unit will receive equivalent dementia care education and training as well as staff support (please refer to NCT# 04179721 for more details on this aim).
  Arms: The attention control condition

SUMMARY:
Persons with Alzheimer's Disease and Related Dementias (ADRD) account for 3.2 million hospital admissions per year and have over three times more hospitalizations than those without cognitive impairment, yet hospital caregivers (HCGs) are ill-prepared to manage patients with ADRD with less than 5% reporting mandatory dementia care training. Three-quarters of hospitalized persons with ADRD display Behavioral and Psychological Symptoms of Dementia (BPSD) associated with functional and cognitive decline, increased resource consumption, institutionalization, premature death, and caregiver burden. The overall objective is to test the preliminary efficacy of an innovative model of care, PES-4-BPSD, for reducing BPSD by empowering Patient Engagement Specialists (PES) to deliver dementia care for acutely-ill patients with ADRD. Traditionally, mental health assistants with training in crisis-prevention techniques provide care to psychiatric patients. On the intervention unit, these mental health assistants, as PES, purposefully engage patients with BPSD. In the pilot study, investigators found patients with cognitive impairment admitted to the PES unit were significantly less likely to require constant observation, chemical and physical restraints, suggesting improved management of BPSD. The central hypothesis is that PES-4-BPSD will improve the ability of PES to create an "enabling" milieu that addresses factors leading to BPSD and improves the experience of hospital caregivers. Guided by a social-ecological framework, PES-4-BPSD incorporates dementia education and training, environmental modifications-cohorting, increased staffing-PES, and staff support. The investigators' multidisciplinary research team is well-positioned to accomplish the following: Aim 1) Determine the preliminary efficacy of PES-4-BPSD for reducing BPSD during hospitalization, and Aim 2) Evaluate whether dementia care training improves the perceived ability of PES staff (intervention) and nurse assistant staff (control) to care for hospitalized persons with ADRD. For Aim 1, investigators will conduct a non-randomized preliminary efficacy trial of the PES-4-BPSD intervention enrolling N=158 patients (79 control, 79 intervention). The primary outcome will be presence of BPSD during hospitalization using the Neuropsychiatric Inventory-Questionnaire (NPI-Q). In Aim 2, investigators will use survey methodology in a repeated measures design to evaluate within and between-group differences in attitudes, experience, and satisfaction toward managing patients with ADRD. Measures will be completed at baseline (T1), immediately following training (T2), and at the end of the intervention period (T3). This proposal will be the first to study an innovative model of care utilizing PES as specialized hospital caregivers for reducing BPSD in the hospital setting. The investigators' findings will lay the essential groundwork for a multi-site trial of PES-4-BPSD and inform the development of a program that can be easily implemented in other hospitals.

DETAILED DESCRIPTION:
Prior to patient recruitment, a 3 month dementia training program will be implemented on both the intervention and control units. On the intervention unit, training will target the Patient Engagement Specialists (PES) and on the control to the nurse assistants (please refer to NCT# 04179721 for more details on this aim). Following the implementation of the dementia care training, eligible patients will be offered the opportunity to participate in the study. A research coordinator will offer the information and opportunity to participate to the patient's lawful caregiver. The signed consent forms will be stored in secured file cabinets. Once a participant has been enrolled in the study, demographic information will be obtained from the electronic medical records (EMR) and verified by Family Caregiver (FCG), including: age, gender, race/ethnicity, marital status, education, work status, current living situation, medical comorbidities, and reason for admission. A member of the research team will conduct a short interview with the FCG to verify patient background information and obtain baseline (1 month prior to admission) functional status (Barthel Index), dementia severity cognitive (Clinical Dementia Rating Scale)(5 stages of severity: no 0, questionable 0.5, mild 1, moderate 2, and severe 3), and behavioral symptoms using the Neuropsychiatric Inventory-Clinical version NPI-C.

A member of the research team will then complete daily NPI-Qs to determine the number of behaviors and symptoms for each patient on a daily basis. The data collector will use a multimodal approach drawing from electronic medical record (EMR) notes and interviews with nursing staff regarding the patient's behavior and treatment over the past 24 hours. Delirium will be assessed daily by the research coordinator using same multimodal approach and during the time of NPI observation. A final EMR chart review will be conducted collecting information such as length of stay, discharge disposition, in-hospital mortality as well as total usage practices for management of BPSD: use of special observation (1:1 or enhanced), restraints, psychoactive medications, psychiatric evaluation. Within 48 hours of discharge, family caregivers will be interviewed regarding satisfaction with care using the Carer Questionnaire Data from the National Audit of Dementia Round 3.

ELIGIBILITY:
Inclusion criteria:

* Patients who have an acute medical admission to either the control unit (Geriatric Care Model) or intervention unit (PES-4-BPSD).
* Patients age 65 and above
* Documentation of dementia in the medical record (based on the International Classification of Diseases, Ninth and Tenth Revision codes [ICD-9 and ICD-10])
* AD8 score of 2 or greater (obtained from the family caregiver [FCG])

Exclusion Criteria:

* Patients who are known to be terminally ill and/or receiving hospice or surgery
* Patients with a length of stay of less than 48 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liron Sinvani, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Long Island Jewish Medical Center, Glen Oaks, New York
  - North Shore University Hospital, Manhasset, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sampson EL, White N, Leurent B, Scott S, Lord K, Round J, Jones L. Behavioural and psychiatric symptoms in people with dementia admitted to the acute hospital: prospective cohort study. Br J Psychiatry. 2014 Sep;205(3):189-96. doi: 10.1192/bjp.bp.113.130948. Epub 2014 Jul 24. PMID 25061120
- [Background] Hessler JB, Schaufele M, Hendlmeier I, Junge MN, Leonhardt S, Weber J, Bickel H. Behavioural and psychological symptoms in general hospital patients with dementia, distress for nursing staff and complications in care: results of the General Hospital Study. Epidemiol Psychiatr Sci. 2018 Jun;27(3):278-287. doi: 10.1017/S2045796016001098. Epub 2017 Jan 9. PMID 28065176
- [Background] Astrom S, Nilsson M, Norberg A, Sandman PO, Winblad B. Staff burnout in dementia care--relations to empathy and attitudes. Int J Nurs Stud. 1991;28(1):65-75. doi: 10.1016/0020-7489(91)90051-4. PMID 1856035
- [Background] Dewing J, Dijk S. What is the current state of care for older people with dementia in general hospitals? A literature review. Dementia (London). 2016 Jan;15(1):106-24. doi: 10.1177/1471301213520172. Epub 2014 Jan 23. PMID 24459188
- [Background] Lintern TC. Quality in dementia care: evaluating staff attitudes and behaviour. [PhD Thesis]. Prifysgol Bangor University; 2001
- [Background] Scerri A, Innes A, Scerri C. Dementia training programmes for staff working in general hospital settings - a systematic review of the literature. Aging Ment Health. 2017 Aug;21(8):783-796. doi: 10.1080/13607863.2016.1231170. Epub 2016 Sep 23. PMID 27662075
- [Result] Sinvani L, Warner-Cohen J, Strunk A, Halbert T, Harisingani R, Mulvany C, Qiu M, Kozikowski A, Patel V, Liberman T, Carney M, Pekmezaris R, Wolf-Klein G, Karlin-Zysman C. A Multicomponent Model to Improve Hospital Care of Older Adults with Cognitive Impairment: A Propensity Score-Matched Analysis. J Am Geriatr Soc. 2018 Sep;66(9):1700-1707. doi: 10.1111/jgs.15452. Epub 2018 Aug 11. PMID 30098015
- See also: Please refer to NCT# 04179721 for more details on Aim 2: Hospital Caregivers — https://clinicaltrials.gov/ct2/show/NCT04179721

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Started | 79 | 79
Completed | 79 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.5 (8.44) | 86.9 (7.48) | 85.2 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 31 | 27 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 16
  Not Hispanic or Latino | 72 | 66 | 138
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 9 | 36
  White | 34 | 59 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Marital Status [Count of Participants; unit: Participants]
  Married/Domestic Partnership | 28 | 26 | 54
  Divorced | 8 | 10 | 18
  Separated | 3 | 1 | 4
  Widowed | 35 | 40 | 75
  Single/Never Married | 5 | 2 | 7
Education [Count of Participants; unit: Participants]
  Less than a high school diploma | 18 | 17 | 35
  High school degree or equivalent | 34 | 33 | 67
  Associates degree (e.g., AA, AS) | 6 | 4 | 10
  Bachelors degree (e.g. BA, BS) | 12 | 7 | 19
  Masters degree (e.g. MA, MS) | 4 | 10 | 14
  Doctorate (e.g. PhD, PsyD) | 0 | 4 | 4
  Other | 5 | 4 | 9
Residence [Count of Participants; unit: Participants]
  Still in own home | 47 | 49 | 96
  Caregivers home | 25 | 9 | 34
  Assisted-living facility | 5 | 12 | 17
  Independent living | 1 | 1 | 2
  Nursing home | 0 | 8 | 8
  Other | 1 | 0 | 1
Previous history of dementia [Count of Participants; unit: Participants]
  Yes | 57 | 70 | 127
  No | 22 | 9 | 31
Charlson Comorbidity Index [Mean (Standard Deviation); unit: score on a scale] — The Charlson Comorbidity Index is a marker of baseline comorbid disease and is based on the presence and severity of 19 comorbidities. Age-adjusted results range from all participants range from 2 - 39, with higher scores indicating greater likelihood of mortality.
  score on a scale | 8.09 (2.66) | 8.77 (2.65) | 8.43 (2.67)
Clinical Dementia Rating Worksheet final score [Count of Participants; unit: Participants]
  0 - No Impairment | 0 | 0 | 0
  0.5 - Questionable Impairment | 3 | 9 | 12
  1 - Mild Impairment | 13 | 12 | 25
  2 - Moderate Impairment | 30 | 21 | 51
  3 - Severe Impairment | 33 | 37 | 70
Baseline Neuropsychiatric inventory questionnaire [Mean (Standard Deviation); unit: score on a scale] — The Neuropsychiatric Inventory Questionnaire (NPI-Q) is a validated tool with 12 behavioral domains for the assessment of neuropsychiatric symptomology designed for completion by caregivers of patients with Alzheimer's Disease and Related Dementias. The tool asks the interviewee to rate each symptom, if present, as mild, moderate, or severe. Total scores range from 0-36 with higher scores indicating greater prominence of dementia symptoms.
  score on a scale | 15.8 (7.49) | 10.5 (6.60) | 13.1 (7.51)

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychiatric Inventory Questionnaire Average Score During Hospital Admission
Description: The Neuropsychiatric Inventory Questionnaire (NPI-Q) is a validated tool with 12 behavioral domains for the assessment of neuropsychiatric symptomology designed for completion by caregivers of patients with Alzheimer's Disease and Related Dementias. The tool asks the interviewee to rate each symptom, if present, as mild, moderate, or severe. Total scores range from 0-36 with higher scores indicating greater prominence of dementia symptoms. A Research Coordinator (RC) will utilize a multimodal approach, consisting of daily NPI-Q interviews with Hospital Caregivers and daily reviews of the patient's medical record, to provide a daily assessment of the 12 NPI-Q domains during hospitalization. Upon discharge, the average of each patient's daily NPI-Q total scores will be calculated, and this average will serve as the primary outcome.
Time Frame: Participant length of stay varies, median of 7 days; will be assessed for 1 year duration of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 79 | 79
score on a scale | 5.36 (4.64) | 3.87 (3.37)

2. Secondary Outcome: Length of Stay
Description: Collected via chart review.
Time Frame: Participant length of stay varies, median of 7 days; will be assessed for 1 year duration of study
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 79 | 79
days | 7.00 [6.40 to 8.14] | 7.86 [5.88 to 9.8]

3. Secondary Outcome: Practices for the Management of BPSD
Description: Collected via chart review. Practices include orders placed for special observation (1:1 or enhanced), restraints, psychoactive medications, psychiatric evaluation, as well as adverse events (falls). Orders for constant observation are reported below.
Time Frame: Outcomes vary by participant; will be assessed through duration of study for 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 79 | 79
Participants | 17 | 15

4. Secondary Outcome: Family Caregiver (FCG) Satisfaction
Description: FCGs will be interviewed by research coordinator with a one-time telephone survey within 48 hours of discharge using the UK National Audit of Dementia Round 3, Caregiver Questionnaire. The survey consists of 10 items assessing perceptions of hospital quality of care provided by hospital staff. Responses of "Excellent" to the primary question assessed, "overall, how would you rate the care received by your loved one during their hospital stay?" is reported.
Time Frame: Collected within 48 hours of hospital discharge for the 1-year study duration
Measure: Count of Participants; unit: Participants
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 79 | 79
Participants | 34 | 26

ADVERSE EVENTS:
Time Frame: Length of inpatient stay (median of 7 days) through 48 hours following hospital discharge; will be assessed for 1 year duration of study
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
All-Cause Mortality (participants affected / at risk) | 0/79 | 2/79
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/79
Other Adverse Events (participants affected / at risk) | 0/79 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04481568/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04481568/ICF_001.pdf